CLINICAL TRIAL: NCT07222150
Title: Unity VCS: A Comparison Study Evaluating Corneal Clarity and Thickness at Day 1 and Day 8 Post Op
Brief Title: Unity VCS: A Comparison Study Evaluating Corneal Clarity and Thickness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Metrolina Eye Associates, PLLC (Other)
Collaborators: Alcon, a Novartis Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IIT# 98711335; IM-25-02 (Other: Advarra IRB)
Record Dates: First submitted 2025-10-13; First posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Cataract
Keywords: Cataract Surgery; Phacoemulsification
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Intervention Model Description: Prospective, two-surgeon, randomized, paired-eye study; patients undergoing sequential, uncomplicated bilateral phacoemulsification using Unity VCS 4D phaco with intraocular IOP ≤ 28mmHg (low IOP) in one eye and with IOP ≥ 65mmHg (high IOP) in the other eye usingCenturion Vision System with Ozil.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Unity VCS (Active Comparator): Cataract surgery with Unity VCS
  Interventions: Device: Cataract surgery with Unity VCS; Device: Cataract surgery with Centurion with Ozil
- Centurion with Ozil (Active Comparator): Cataract surgery with Centurion with Ozil
  Interventions: Device: Cataract surgery with Unity VCS; Device: Cataract surgery with Centurion with Ozil

INTERVENTIONS:
Device: Cataract surgery with Unity VCS — Standard cataract surgery
Device: Cataract surgery with Centurion with Ozil — Standard cataract surgery

SUMMARY:
Phacoemulsification (cataract surgery) is usually performed while temporarily increasing the pressure inside the eye. The purpose of this study is to see if maintaining different pressure levels inside the eye during this procedure results in fewer side effects and better vision shortly after the surgery. Cataract surgery will be performed using Unity VCS at a lower IOP in one eye compared to traditional IOP with Centurion Vision System with Ozil in the other eye. Both of which are approved by the United States Food and Drug Administration (FDA) and used per label.

DETAILED DESCRIPTION:
Study patients will undergo sequential bilateral cataract surgery with the same cataract grade in both eyes. Both surgeries will be completed within one week of each other.

The first surgical eye will be randomly assigned (like the flip of a coin). Study patients will have surgery performed with the Alcon Unity VCS system using 4D. The second eye will undergo surgery a week later with Alcon Centurion Vision System (VCS) with Ozil. Surgery with the Unity VCS arm will be performed with a lower IOP setting (less than 40). Surgery with the Centurion with Ozil arm will be performed with a higher IOP setting (greater or equal 60).

Participation in the study is expected to take one month.

ELIGIBILITY:
Inclusion Criteria:

* Cataracts

Exclusion Criteria:

* Glaucoma, cornea disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Central corneal thickness (CCT) | Pre-operative, Post-operative day #1, Post-operative day #8 for each arm of the study
  Measurement of post-operative CCT pre and post-operatively with Pentacam

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Mac, MD, Principal Investigator — Metrolina Eye Associates
Locations (1):
- Metrolina Eye Associates, Matthews, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Only summary data will be published comparing the two study arms.

REFERENCES:
- [Background] Liu Y, Hong J, Chen X. Comparisons of the clinical outcomes of Centurion(R) active fluidics system with a low IOP setting and gravity fluidics system with a normal IOP setting for cataract patients with low corneal endothelial cell density. Front Med (Lausanne). 2023 Nov 23;10:1294808. doi: 10.3389/fmed.2023.1294808. eCollection 2023. PMID 38076276
- [Background] Spaulding J, Hall B. Efficiency of phacoemulsification handpieces with high and low intraocular pressure settings. J Cataract Refract Surg. 2025 Mar 1;51(3):218-221. doi: 10.1097/j.jcrs.0000000000001581. PMID 39602355
- [Background] Rauen MP, Joiner H, Kohler RA, O'Connor S. Phacoemulsification using an active fluidics system at physiologic vs high intraocular pressure: impact on anterior and posterior segment physiology. J Cataract Refract Surg. 2024 Aug 1;50(8):822-827. doi: 10.1097/j.jcrs.0000000000001457. PMID 38595209

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT07222150/Prot_SAP_000.pdf